CLINICAL TRIAL: NCT02868359
Title: PATIENT-REPORTED-OUTCOMES IN CHRONIC CERVICAL PAIN PATIENTS WITH ACCOMPANYING UPPER LIMB RADIATING PAIN (NEUROPATHIC COMPONENT) TREATED WITH PREGABALIN IN PRIMARY CARE SETTINGS
Brief Title: PROs in Chronic Cervical Pain Patients With Accompanying Upper Limb Radiating Pain Treated With Pregabalin
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081354
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2019-01

CONDITIONS: Cervical Pain; Neuropathic Pain; Radiating Pain
MeSH Terms: conditions — Neck Pain; Neuralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregabalin / Other analgesics: Patients will be treated for 8 weeks with pregabalin in primary care: no intervention
  Interventions: Other: No Intervention
- Other analgesics: Patients will be treated for 8 weeks with other analgesics in usual care: no intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — The study is observational.

SUMMARY:
The purpose of this study is to evaluate the effect of pregabalin on patient reported outcomes compared with conventional analgesic care in chronic cervical pain patients with accompanying upper limb radiating pain (neuropathic component) treated in primary care settings under routine clinical practice.

DETAILED DESCRIPTION:
Rational and background:

Cervical pain with upper limb radiating pain(neuropathic component), such as cervical spondylosis radiculopathy or cervical spondylotic myelopathy, is one of the typical and common neuropathic pain. However, in Japan, large number of those patients are treated with NSAIDs without adequately assessing the cause of pain, despite that α2δ ligand, SNRI (Serotonin and Norepinephrine Reuptake Inhibitors ), and TCA (Tricyclic Antidepressants) are recommended in the clinical guidelines for neuropathic pain. Therefore, treatment satisfaction of these patients is low. This is currently a major issue in treatment for cervical pain with neuropathic component in Japan. In fact, our previous study which assessed the effect of pregabalin in low back pain patients with radiculopathy suggested that the selection of appropriate analgesics according to the cause of pain improved pain related sleep interference, pain and function. However, there are a few reports with regard to effect of pregabalin in cervical pain patients with neuropathic component. Therefore, we propose to conduct an observational study in order to assess the effects of pregabalin in cervical radiculopathy, when added to routine clinical care. The present study can encourage an understanding of the necessary of assessing cause of the pain, and treating with appropriate analgesics.

Research objectives :

To evaluate the effect of pregabalin comparing with the conventional analgesic care in chronic cervical pain patients with accompanying upper limb radiating pain(neuropathic component) treated in primary care settings under routine clinical practice.

Study design:

This is an 8-week, multicenter prospective non-interventional observational study. Subjects who have chronic cervical radiating pain patients with accompanying upper limb radiating pain (with a neuropathic component) and meet all other entry criteria are enrolled at baseline in the duration of study. Study arms are pregabalin with or without usual care vs. usual care (mono/combo therapy). The usual care are assumed NSAIDs, Antidepressants, weak opioids, acetaminophen etc.

The analgesic treatment is determined by the clinical judgment of the physician in charge of patient management. This therapeutic choice is not related to the decision to take part in the study. All enrolled subjects will be received with analgesic treatment. The study requires 3 visits at least, baseline/enrollment visit, Week 4 visit and Week 8 visit (or discontinuation).

ELIGIBILITY:
Inclusion Criteria:

Subject who received the enough study information and signed informed consent form.

Subject who had chronic pain with accompanying radiating pain to the superior limb beyond the elbow.

Subject is male or female patient ≧20 years old. Subject who reported neck pain with accompanying radiating pain to superior limb (12 weeks or greater in duration at Visit 0).

Subject who is refractory to previous analgesics for 12 weeks and more. Subject who is able and willing to complete all study related assessment tools and complied with scheduled clinic visits and clinical study procedures.

Subject whose pain NRS ≧5 and PRSIS ≧1 at baseline (based on recall over the past week).

Exclusion Criteria:

Subject who, in the opinion of the investigator, was not likely to complete the trial for whatever reason.

Subject who was treated with Pregabalin within the past 12 weeks (on baseline). Subject who has been regularly treated cervical pain with nerve blocks (such as stellate ganglion block, epidural block, radicular block and trigger point injection etc.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic cervical pain patients with accompanying upper limb radiating pain (neuropathic component) treated with pregabalin or other analgesics
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Change From Baseline at 8 weeks in Pain Related Sleep Interference Scale (PRSIS - Past Week Recall) | Baseline, Visit 2 (week 4), Final visit (week 8 or discontinuation)
  The Pain Related Sleep Interference Scale (past week recall) consists of an 11-point numeric rating scale (NRS) ranging from 0 (pain did not interfere with sleep) to 10 (pain completely interfered with sleep). Subjects are to describe how their pain has interfered with their sleep during the past week by choosing the appropriate number between 0 and 10.

SECONDARY OUTCOMES:
Change From Baseline in Neck Disability Index (NDI) | Baseline, Visit 2 (week 4), Final visit (week 8 or discontinuation)
  The Neck Disability Index (NDI) is an index of how well patients with cervical pain are able to function with regard to daily activities. The score for the index ranges from 0 to 50 with a lower score indicating better function. In the event that a patient has used rescue medication within 12 hours of the clinic visit, the patient should respond to the questions based on their functional ability in the 24 hour period just preceding the use of rescue medication.
Change From Baseline in Pain Numeric Rating Scale (Pain NRS - past week recall) | Baseline, Visit 2 (week 4), Final visit (week 8 or discontinuation)
  The Pain NRS (past week recall) consists of an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain). Subjects are asked to describe their average pain during the past week by choosing the appropriate number between 0 and 10.
Change From Baseline in Euro Qol- 5 Dimensions -5 Level (EQ-5D-5L)-QOL-Score- | Baseline, Visit 2 (week 4), Final visit (week 8 or discontinuation)
  The EQ-5D-5L is a copyrighted, subject-completed questionnaire designed to assess health-related quality of life in terms of a single index value or utility score. There are two components to the EQ-5D-5L: A Health State Profile and a Visual Analogue Scale (VAS). Recent guidance suggests that the Health State Profile and VAS should be administered together.
  The Health State Profile is designed to record the subject's level of current health for five domains comprising a health profile: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Responses from the five domains are used to calculate a single utility index value.
Change From Baseline in Euro Qol- 5 Dimensions -5 Level (EQ-5D-5L)-Visual Analogue Scale - | Baseline, Visit 2 (week 4), Final visit (week 8 or discontinuation)
  The EQ-5D-5L is a copyrighted, subject-completed questionnaire designed to assess health-related quality of life in terms of a single index value or utility score. There are two components to the EQ-5D-5L: A Health State Profile and a Visual Analogue Scale (VAS). Recent guidance suggests that the Health State Profile and VAS should be administered together.
  The Visual Analogue Scale (VAS) is designed to rate the subject's current health state on a scale from 0 to 100 where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Clinical Global Impression of Change (CGIC) | Final visit (week 8 or discontinuation)
  The CGIC assessment includes one question (1-7 scale) inquiring about the subject's improvement considering their current disease state.
Patient Global Impression of Change (PGIC) | Final visit (week 8 or discontinuation)
  The PGIC is a subject-rated instrument that measures change in the subject's overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse).
Work Productivity and Activity Impairment Questionnaire: (WPAI: GH) | Final visit (week 8 or discontinuation)
  The WPAI: GH is a self-administered questionnaire that measures the effect of general health and symptom severity on work productivity and regular activities. Unlike general health or disease-specific measures, the WPAI:GH assesses function-related endpoints to allow a measure of the economic impact of relative differences in either the safety or efficacy of therapeutic endpoints. In this study, the WPAI: GH will measure the effect of the patient's chronic cervical pain with accompanying upper limb pain (neuropathic component) on work productivity and regular activities.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Japan (33):
  - Satoh Orthopaedic Clinic, Ichikawa, Chiba
  - Shiraishi Orthopaedic Clinic, Ichikawa, Chiba
  - Clinic for Sports Medicine and Nutrition, Fukuoka, Fukuoka
  - Seiwa Orthopedics Surgery Internal Medicine, Fukuoka, Fukuoka
  - Kiheikai Yoh Orthopedic Clinic, Fukuoka, Fukuoka
  - Chihaya Hospital, Fukuoka, Fukuoka
  - Fukuoka Mirai Hospital, Higashi-ku,Fukuoka, Fukuoka
  - Shin Komonji Hospital, Kitakyusyu-shi, Fukuoka
  - Fukushima Daiichi Hospital, Fukushima, Fukushima
  - Takasaki Pain Clinic, Takasaki-shi, Gunma
  - Miyanomori Memorial Hospital, Sapporo, Hokkaido
  - Oomuro Orthopedic Clinic, Himeji-shi, Hyōgo
  - Oonishi Medical Clinic, Kako-gun, Hyōgo
  - Watanabe Orthopaedic Clinic, Kobe, Hyōgo
  - Fujisawa Shonandai Hospital, Fujisawa-shi, Kanagawa
  - Ando Orthopaedics Hospital, Kawasakishi, Kanagawa
  - General Sagami Kosei Hospital, Sagamiharashi, Kanagawa
  - Arai Orthopaedic Clinic, Saitama, Kanagawa
  - Saitoh Orthopedic Sports Clinic, Yamato-shi, Kanagawa
  - Ageo Medical Clinic, Ageo, Saitama
  - Nakaicho Clinic, Adachi City, Tokyo
  - Kyobashi Orthopaedic Clinic, Chūō, Tokyo
  - Morishima Clinic, Edogawa City, Tokyo
  - Shinkoiwa Ekimae Sogo Clinic, Katsushika-ku, Tokyo
  - Meguro Seikeigeka Naika, Meguro City, Tokyo
  - Meguro Yuai Clinic, Meguro City, Tokyo
  - Takemoto Orthopaedic Clinic, Ohta, Tokyo
  - Ohimachi Orthopaedic Clinic, Shinagawa, Tokyo
  - Shinjuku Research Park Clinic, Shinnzyuku, Tokyo
  - Kouenji Orthopedic Clinic, Suginami, Tokyo
  - Daido Hospital, Toshima City, Tokyo
  - Saga-ken Medical Center Koseikan, Saga
  - Tokyo Rheumatism Pain Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Taguchi T, Nozawa K, Parsons B, Yoshiyama T, Ebata N, Igarashi A, Fujii K. Effectiveness of pregabalin for treatment of chronic cervical radiculopathy with upper limb radiating pain: an 8-week, multicenter prospective observational study in Japanese primary care settings. J Pain Res. 2019 May 3;12:1411-1424. doi: 10.2147/JPR.S191906. eCollection 2019. PMID 31118759
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081354&StudyName=Patient-reported-outcomes+In+Chronic+Cervical+Pain+Patients+With+Accompanying+Upper+Limb+Radiating+Pain+%28neuropathic+Component%29+Treated+With+Pregabalin+In+Primary+Care+Settings